CLINICAL TRIAL: NCT02382432
Title: Safety and Efficacy of Dexmedetomidine in Treating Post Spinal Anesthesia Shivering: A Clinically Controlled Dose-finding Study.
Brief Title: Dexmedetomidine in Post Spinal Anesthesia Shivering
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, Assistant professor in anesthesia department, faculty of medicine, Assiut university, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00008718
Record Dates: First submitted 2015-02-25; First posted 2015-03-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Shivering Caused by Spinal Anesthesia
Keywords: Anesthesia; dexmedetomidine; pethidine; shivering; spinal
MeSH Terms: interventions — Meperidine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pethidine 0.4mg/kg iv (Active Comparator): interventional: Pethidine 0.4mg/kg intravenous bolus once to be repeated if shivering incompletely abolished.
  Interventions: Drug: Pethidine 0.4mg/kg
- DEX. I (Active Comparator): Interventional:Dexmedetomidine (Precedex) 0.5µg/kg intravenous bolus once to be repeated if shivering incompletely abolished.
  Interventions: Drug: Dexmedetomidine
- DEX. II (Active Comparator): Interventional: Dexmedetomidine (PRECEDEX) 0.3µg/kg intravenous bolus given once to be repeated if shivering incompletely abolished.
  Interventions: Drug: Dexmedetomidine
- DEX III (Active Comparator): Interventional: Dexmedetomidine (PRECEDEX) 0.2µg/kg intravenous bolus given once to be repeated if shivering incompletely abolished.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Pethidine 0.4mg/kg — 2ml intravenous bolus slowly injected in 2minutes.
  Other Names: Meperidine
  Arms: Pethidine 0.4mg/kg iv
Drug: Dexmedetomidine — 2ml intravenous bolus slowly injected in 2minutes
  Other Names: Precedex
  Arms: DEX III; DEX. I; DEX. II

SUMMARY:
This study evaluated the effect of dexmedetomidine iv in three different doses in the treatment of shivering in patients undergoing minor elective abdominal surgery under spinal anesthesia, in comparison with intravenous pethidine.

DETAILED DESCRIPTION:
Among the pharmacological agents used in treatment of shivering, pethidine (meperidine) has been shown to be one of the most effective treatments.The α-2 receptor agonists are another important class of anti-shivering drugs that, unlike meperidine, produce little respiratory depression.

Dexmedetomidine is a highly selective α-2 adrenoceptor agonist with potent effects on the central nervous system . Intravenous dexmedetomidine reduces both the vasoconstriction and shivering thresholds . Clinical studies had demonstrated the efficacy of dexmedetomidine in prevention of shivering . Few clinical trials investigated its efficacy in treatment of established shivering. The optimum dose for shivering control with the least hemodynamic derangements is still under research.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist class I or II scheduled for elective minor lower abdominal operations under spinal anesthesia for an anticipated duration of >60 and <180 min. (e.g. inguinal herniorRaphy, umbilical hernia repair) who developed shivering during the intra or postoperative period

Exclusion Criteria:

* Patients with BMI>30 kg /m2
* Initial body temperature >38 C or <36 C and those with a history of convulsions
* Multiple allergies
* Thyroid disease
* Parkinson's disease
* Dysautonomia
* Raynaud's syndrome
* Hypertension
* Coronary artery disease or other cardio-respiratory or neuromuscular pathology
* Middle ear pathology
* A known history of alcohol use
* Treatment with sedative hypnotic agents or vasodilators
* Having contraindications to spinal anesthesia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Shivering response rate (%) | 10 minutes
  complete cessation of shivering activity within 10 minutes after study drug injection

SECONDARY OUTCOMES:
Systolic blood pressure | 6 hours after study drug injection
  find for systolic hypotension, hypertension
sedation | 6 hours after study drug injection
  using an Observer's Assessment of Alertness/Sedation Scale (OAA/SS) (where 5 = Responds readily to name spoken in normal tone, 4 = Lethargic response to name spoken in normal tone, 3 = Responds only after name is spoken loudly and/or repeatedly, 2 = Responds only after mild prodding or shaking, 1 = Does not respond to mild prodding or shaking).
peripheral arterial saturation | 6 hours after study drug injection
  find for hypoxia
diastolic blood pressure | 6 hours after study drug injection
  find for diastolic hypertension or hypotension
Postoperative adverse events | 24 hours postoperative
  postoperative nausea and vomiting, urine retention, post dural puncture headache ect.

OTHER OUTCOMES:
heart rate | 6 hours after study drug injection
  find for bradycardia or tachycardia

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdel-Ghaffar, MD, Principal Investigator — assistant professor in anesthesia, faculty of medicine, Assiut university, Assiut, Egypt
Locations (1):
- Assiut university hospital, Assiut, Egypt, Asyut, Assiut Governorate, Egypt

REFERENCES:
- [Derived] Abdel-Ghaffar HS, Mohamed SA, Fares KM, Osman MA. Safety and Efficacy of Dexmedetomidine in Treating Post Spinal Anesthesia Shivering: A Randomized Clinically Controlled Dose-Finding Trial. Pain Physician. 2016 May;19(4):243-53. PMID 27228512